CLINICAL TRIAL: NCT01438866
Title: The Effectiveness of Sealants in Prevention of Occlusal Caries on Primary Molars
Brief Title: Use of Fissure Sealants on Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, Sisko Honkala, Associate Professor, Kuwait University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DD03/10
Record Dates: First submitted 2011-09-18; First posted 2011-09-22 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2012-10

CONDITIONS: Dental Caries
Keywords: Dental caries; Fissure sealant; Fluoride varnish; Primary molar
MeSH Terms: conditions — Dental Caries | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preventing occlusal caries (Experimental): Comparing preventing effect of fissure sealants vs. fluoride varnish
  Interventions: Other: Fissure sealant; Other: Fissure sealants and fluoride varnish

INTERVENTIONS:
Other: Fissure sealant — Preventing dental caries in primary molars by applying fissure sealants and fluoride varnish, and comparing caries preventive effect of sealants with fluoride varnish.
  Other Names: Brand name: Clinpro™ Sealant; Produced by: 3M ESPE; www.3MESPE.com/PrventiveCare; Brand name: DuraShield® 5% Sodium Fluoride Varnish; Produced by: Sultan Dental Products; www.sultandental.com
Other: Fissure sealants and fluoride varnish — Comparing preventive effect of fissure sealants and fluoride varnish on occlusal surfaces of primary molars
  Other Names: ClinproTM (3M ESPE); DuraShield® (Sultan Healthcare)

SUMMARY:
Sealants have been shown to be the most effective caries preventive measure in permanent dentition. Sealants of the primary molars soon after they erupt would reduce the total caries experience of the primary teeth of the children and could possibly also postpone the caries process in the permanent dentition.

The aim of this study is to measure the caries preventive effect of sealants in primary molars. The specific objectives are: 1) to compare the number of new caries experience teeth and surfaces among the intervention group of 4-years old pre-school children during the 1 year follow-up period, 2) to compare the preventive effect of sealants with fluoride varnish on the caries experience on the occlusal surfaces of the primary molars and on the total caries experience of all the primary and permanent teeth, 3) to test the feasibility of the sealant program in one kindergarten in Kuwait city.

ELIGIBILITY:
Inclusion Criteria:

* positive written informed consent received from parents

Exclusion Criteria:

* if caries lesions in primary molars are so extensive that restorative treatment is needed

Ages: 42 Months to 52 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of healthy occlusal tooth surfaces of primary molars | up to 1 year
  Outcome will be measured by a clinical examination (dental caries status/ICDAS) one year after the fissure sealants and fluoride varnish have been applied. When a child has intact occlusal surfaces on primary molars in the baseline examination, s/he will get a fissure sealant on the other side of the mouth and fluoride varnish on the other side.

SECONDARY OUTCOMES:
Number of healthy occlusal tooth surfaces after application of fissure sealants versus fluoride varnish | up to 1 year
  Outcome will be measured by a clinical examination (dental caries status/ICDAS)one year after the fissure sealants and fluoride varnish have been applied. The effectiveness of these two preventive treatment will be compared, i.e. how many occlusal surfaces of primary molars stayed caries free with the sealant application vs. fluoride varnish application.

CONTACTS AND LOCATIONS:
Overall Officials: Sisko L Honkala, DDS, PhD, Principal Investigator — Faculty of Dentistry, Kuwait University
Locations (1):
- Kindergarten, Kuwait City, Hawally, Kuwait

REFERENCES:
- See also: Related Info — http://www.hsc.edu.kw/fod/